CLINICAL TRIAL: NCT05046678
Title: Effects of Smoking on Saliva MicroRNAs Before and After Non-Surgical Periodontal Therapy in Patients With Periodontal Disease
Brief Title: miRNAs in Periodontal Disease
Status: Completed | Type: Observational
Sponsor: Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, Figen Öngöz Dede, T.C. ORDU ÜNİVERSİTESİ, Bulent Ecevit University
Other Study IDs: 318S106
Record Dates: First submitted 2021-09-13; First posted 2021-09-16 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Periodontal Diseases; Periodontitis; Gingivitis
MeSH Terms: conditions — Periodontal Diseases; Periodontitis; Gingivitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Weeks
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Control: Periodontally healthy, non-smoking
  Interventions: Diagnostic Test: Smokers with periodontally healthy; Diagnostic Test: Non-smokers with gingivitis; Diagnostic Test: Smokers with gingivitis; Diagnostic Test: Non-smokers with periodontitis; Diagnostic Test: Smokers with periodontitis
- Smokers with periodontally healthy: Periodontally healthy, smoking
  Interventions: Diagnostic Test: Control; Diagnostic Test: Non-smokers with gingivitis; Diagnostic Test: Smokers with gingivitis; Diagnostic Test: Non-smokers with periodontitis; Diagnostic Test: Smokers with periodontitis
- Non-smokers with gingivitis: Gingivitis, non-smoking
  Interventions: Diagnostic Test: Control; Diagnostic Test: Smokers with periodontally healthy; Diagnostic Test: Smokers with gingivitis; Diagnostic Test: Non-smokers with periodontitis; Diagnostic Test: Smokers with periodontitis
- Smokers with gingivitis: Gingivitis, smoking
  Interventions: Diagnostic Test: Control; Diagnostic Test: Smokers with periodontally healthy; Diagnostic Test: Non-smokers with gingivitis; Diagnostic Test: Non-smokers with periodontitis; Diagnostic Test: Smokers with periodontitis
- Non-smokers with periodontitis: Periodontitis, non-smoking
  Interventions: Diagnostic Test: Control; Diagnostic Test: Smokers with periodontally healthy; Diagnostic Test: Non-smokers with gingivitis; Diagnostic Test: Smokers with gingivitis; Diagnostic Test: Smokers with periodontitis
- Smokers with periodontitis: Periodontitis, smoking
  Interventions: Diagnostic Test: Control; Diagnostic Test: Smokers with periodontally healthy; Diagnostic Test: Non-smokers with gingivitis; Diagnostic Test: Smokers with gingivitis; Diagnostic Test: Non-smokers with periodontitis

INTERVENTIONS:
Diagnostic Test: Control — probing pocket depth (PPD)≤ 3 mm (presence of normal gingival sulcus), bleeding on probing (BOP) < 10%, clinical absence of periodontal inflammation, radiological bone loss, and any prior periodontal disease, additionally presence of anatomically intact periodontium and nonsmokers if they had no previous history of smoking
  Groups: Non-smokers with gingivitis; Non-smokers with periodontitis; Smokers with gingivitis; Smokers with periodontally healthy; Smokers with periodontitis
Diagnostic Test: Smokers with periodontally healthy — probing pocket depth (PPD)≤ 3 mm (presence of normal gingival sulcus), bleeding on probing (BOP) < 10%, clinical absence of periodontal inflammation, radiological bone loss, and any prior periodontal disease, additionally presence of anatomically intact periodontium and smokers if they had smoked ≥10 cigarettes/day for ≥5 years
  Groups: Control; Non-smokers with gingivitis; Non-smokers with periodontitis; Smokers with gingivitis; Smokers with periodontitis
Diagnostic Test: Non-smokers with gingivitis — without attachment and alveolar bone loss who had gingival inflammation, PD ≤ 3 mm and BOP > 30% in the full mouth and nonsmokers if they had no previous history of smoking
  Groups: Control; Non-smokers with periodontitis; Smokers with gingivitis; Smokers with periodontally healthy; Smokers with periodontitis
Diagnostic Test: Smokers with gingivitis — without attachment and alveolar bone loss who had gingival inflammation, PD ≤ 3 mm and BOP > 30% in the full mouth and smokers if they had smoked ≥10 cigarettes/day for ≥5 years
  Groups: Control; Non-smokers with gingivitis; Non-smokers with periodontitis; Smokers with periodontally healthy; Smokers with periodontitis
Diagnostic Test: Non-smokers with periodontitis — interdental clinical attachment level (CAL) ≥ 5 mm and PPD ≥ 6 mm on at least two non-adjacent teeth, bone loss involving the middle or apical third of the root radiographically, moderate ridge defect and ≥30% of teeth and nonsmokers if they had no previous history of smoking
  Groups: Control; Non-smokers with gingivitis; Smokers with gingivitis; Smokers with periodontally healthy; Smokers with periodontitis
Diagnostic Test: Smokers with periodontitis — interdental clinical attachment level (CAL) ≥ 5 mm and PPD ≥ 6 mm on at least two non-adjacent teeth, bone loss involving the middle or apical third of the root radiographically, moderate ridge defect and ≥30% of teeth and smokers if they had smoked ≥10 cigarettes/day for ≥5 years
  Groups: Control; Non-smokers with gingivitis; Non-smokers with periodontitis; Smokers with gingivitis; Smokers with periodontally healthy

SUMMARY:
It has been stated that microRNA (miRNA) play an important role in development, homeostasis and immune functions, and abnormal miRNA expression may cause faster disease progression. The aim of this study was to determine miR-203, miR-142-3p, miR-146a, miR-146b, miR-155, miR-29b gene expressions in saliva of the patients with periodontal disease before and after non-surgical periodontal therapy (NSPT) and to evaluate the effect of smoking on these miRNAs. A total of 90 individuals, 30 with periodontitis, 30 with gingivitis, and 30 periodontally healthy (control group), were included. These three groups were divided into subgroups as smoking and non-smoking individuals, with 15 people in each group. NSPT was applied to patients with periodontitis and gingivitis. Saliva samples and clinical parameters were taken from at baseline and repeated 6 weeks after NSPT.

ELIGIBILITY:
Inclusion Criteria:

Have at least 20 natural teeth, excluding third molars. Periodontitis patients had at least two non-adjacent sites per quadrant with probing depth (PD) ≥ 5 mm and clinical attachment level (CAL) ≥ 5 mm with gingival inflammation, and alveolar bone loss affecting >30% of the teeth, as detected on clinical and radiographical examinations.

Gingivitis patients had without attachment and alveolar bone loss who had gingival inflammation, PD ≤ 3 mm and BOP > 30% in the entire mouth Periodontally healthy control group had no sign of gingival inflammation, no PD > 3mm and no evidence of attachment or bone loss

Exclusion Criteria:

History of systemic disease. Regular use of any drugs which can effect the immune system or inflammatory response in the 6 months preceding the start of the study.

Periodontal treatment during last 6 months that could affect periodontal status.

History of radiotherapy or chemotherapy. Current pregnancy, lactation or menopause.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 1. group (Control): Periodontally and systemically healthy and non-smoking
  2. group: Periodontally and systemically healthy and smoking
  3. group: Gingivitis, Systemically healthy and non-smoking
  4. group: Gingivitis, Systemically healthy and smoking
  5. group: Periodontitis, Systemically healthy and non-smoking
  6. group: Periodontitis, Systemically healthy and smoking
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
miRNAs gene expressions in the periodontal disease | baseline
  miR-203, miR-142-3p, miR-146a, miR-146b, miR-155, miR-29b gene expressions in saliva

SECONDARY OUTCOMES:
miRNAs gene expressions in the periodontal disease | baseline and 6 weeks after treatment
  miR-203, miR-142-3p, miR-146a, miR-146b, miR-155, miR-29b gene expressions in saliva before and after non-surgical periodontal treatment

OTHER OUTCOMES:
miRNAs gene expressions in the periodontal disease | baseline and 6 weeks after treatment
  miR-203, miR-142-3p, miR-146a, miR-146b, miR-155, miR-29b gene expressions in saliva of the individials with smokers and nonsmokers

CONTACTS AND LOCATIONS:
Locations (1):
- Ordu University, Ordu, In the USA Or Canada, Please Select..., Turkey (Türkiye)